CLINICAL TRIAL: NCT03861338
Title: An Open-Label Pilot Study of Sublocade as Treatment for Opiate Use Disorder
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Responsible Party: Principal Investigator, John Mariani MD, Research Psychiatrist, New York State Psychiatric Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 7764
Record Dates: First submitted 2019-03-01; First posted 2019-03-04 (Actual); Results first posted 2021-03-09 (Actual); Last update posted 2021-03-09 (Actual); Status verified 2021-02

CONDITIONS: Opioid-use Disorder
Keywords: opioid use disorder, sublocade, buprenorphine
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Sublocade

STUDY DESIGN:
Intervention Model Description: open label pilot for sublocade
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- sublocade (Experimental): Sublocade buprenorphine extended-release (BXR) injection, 300 mg and 100 mg
  Interventions: Drug: Sublocade

INTERVENTIONS:
Drug: Sublocade — The monthly Sublocade buprenorphine extended-release (BXR) injection will be administered in two doses (100 mg and 300 mg). Following a 4 day induction onto oral buprenorphine, the first 300 mg injection of Sublocade will be administered. A second 300 mg Sublocade injection will be administered 1 month later and the third and final monthly injection of 100 mg of Sublocade will be administered 2 months post the successful buprenorphine induction.
  Other Names: buprenorphine extended-release injection

SUMMARY:
The proposed study is a 12-week, open-label pilot study of sublocade (extended-release burprenorphine, BXR) as treatment for opiate use disorder (OUD) testing positive for Highly Potent Synthetic Opioids (HPSO). The investigators plan to enroll 10 participants into the study.

DETAILED DESCRIPTION:
This is an open-label, uncontrolled pilot study. Outpatients seeking treatment for Opiate Use Disorder (OUD) will be screened, and those eligible who are positive for fentanyl analogues at screening will be consented and inducted onto sublingual buprenorphine (target dose 16mg to 24mg). On the fourth day after starting the buprenorphine induction, participants will receive sublocade (BXR) 300mg by subcutaneious injection. Participants will be seen twice per week for urine collection for toxicology and research assessments and will have Medication Management counseling weekly during one of these visits. BXR will be administered monthly and dosing will be according to the FDA prescribing instructions of 300mg for the second dose and 100mg for the third.

ELIGIBILITY:
Inclusion Criteria:

* Individuals between the ages of 18-65
* Voluntarily seeking treatment for opioid use
* Meets current DSM-5 (Diagnostic and Statistical Manual) criteria for Opioid Use Disorder (OUD) as a primary diagnosis, with at least moderate severity
* Test positive for Highly Potent Synthetic Opioids (HPSO) use
* Able to provide informed consent and comply with study procedures

Exclusion Criteria:

* Meets DSM-5 criteria for substance use disorder other than opioid as the primary diagnosis
* Having a comorbid psychiatric diagnosis that might interfere with participation or make participation hazardous, such as an active psychotic disorder or current suicide risk
* Methadone maintenance treatment
* Buprenorphine maintenance treatment
* Known history of allergy, intolerance, or hypersensitivity to candidate medication (buprenorphine)
* Pregnancy, lactation, or failure to use adequate contraceptive methods in female patients, male participants are required to use adequate forms of birth control as the exposure to Sublocade on sperm and subsequent fetal development are not known.
* Unstable medical conditions, which might make participation hazardous such as uncontrolled hypertension (blood pressure >150/100), acute hepatitis, uncontrolled diabetes, or elevated liver function tests (AST (aspartate transaminase) and ALT (alanine aminotransferase) >3 times the upper limit of normal
* Legally mandated to substance use disorder treatment
* Current physiological dependence on alcohol or sedative-hypnotics that would require a medically supervised detoxification-other substance use diagnoses are not exclusionary
* Individuals, who in the clinicians judgment, have a history of failed trial of buprenorphine or sublocade (e.g. history of severe opioid intoxication or overdoses despite adequate adherence to buprenorphine or sublocade), or other features of the history that strongly suggest the patient is not a good candidate for outpatient treatment with buprenorphine.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Mariani, MD, Principal Investigator — New York Psychiatric Institute
Locations (1):
- Substance Treatment Research Service (STARS) of Columbia University, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results published in this report (after de-identification) (text, tables, figures)
Supporting Information: Study Protocol, SAP, ICF
Time Frame: beginning 3 months and ending 5 years after article publication
Access Criteria: to researcher who provides a methodologically sound proposal to achieve aims in the approved proposal

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 10 of the 11 enrolled participants initiated the oral Buprenorphine induction process. 1 participant did not initiate the induction process following consent.
Period: Overall Study
Arm/Group | Sublocade
Started | 10
Completed | 8
Not Completed | 2

BASELINE CHARACTERISTICS:
Population: 10 participants who initiated the induction process
Arm/Group | Sublocade
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.4 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 3
  More than one race | 4
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Sublocade Induction
Description: Number of participants successfully inducted onto Sublocade (BXR)
Time Frame: Study week 1
Measure: Count of Participants; unit: Participants
Arm/Group | Sublocade
Number analyzed (Participants) | 10
Participants | 10

ADVERSE EVENTS:
Time Frame: 12 weeks of study
Arm/Group | Sublocade
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 9/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sublocade (N=10)
opioid withdrawal (General disorders) | 9 (9)
anorexia (Gastrointestinal disorders) | 2 (2)
blurred vision (Eye disorders) | 1 (1)
constipation (Gastrointestinal disorders) | 1 (1)
depression (Psychiatric disorders) | 1 (1)
difficulties with memory (Nervous system disorders) | 1 (1)
fever (General disorders) | 1 (1)
headache (General disorders) | 2 (2)
loss of libido (General disorders) | 1 (1)
tremor (Nervous system disorders) | 1 (1)
increase in weight (Metabolism and nutrition disorders) | 1 (1)
toothache (General disorders) | 1 (1)
cough (Respiratory, thoracic and mediastinal disorders) | 3 (3)
elevated liver functions (Endocrine disorders) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 1 (1)
pharyngitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
sinusitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
injection site pain (Skin and subcutaneous tissue disorders) | 3 (3)
pruritis (Skin and subcutaneous tissue disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2019-02-27): https://cdn.clinicaltrials.gov/large-docs/38/NCT03861338/Prot_000.pdf
  • Statistical Analysis Plan (2019-02-25): https://cdn.clinicaltrials.gov/large-docs/38/NCT03861338/SAP_001.pdf